CLINICAL TRIAL: NCT07030946
Title: The Effectiveness of Multimedia Health Education Interventions in Reducing Surgical Anxiety and Enhancing Care Awareness Among Cataract Surgery Patients
Brief Title: Multimedia Education to Reduce Anxiety and Improve Care Awareness in Cataract Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202500170B0C5001
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Anxiety
Keywords: Self-Care Awareness; Multimedia Health Education; Cataract Surgery; Preoperative Anxiety; Patient Education as Topic; Nursing Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Cataract; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm parallel group trial comparing standard education vs. multimedia education
Who Masked: Participant
Masking Description: This study adopts a randomized experimental research design with two-group repeated measures. A single-blind procedure is implemented, in which patients are blinded to group allocation (patient blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive standard preoperative education, including verbal explanation and printed materials about cataract surgery and postoperative care, provided by the ophthalmologist during the final clinic visit before surgery.
- Multimedia Education Group (Experimental): Participants in the multimedia education group will receive the same standard preoperative education as the control group, plus a 10-minute multimedia video covering the surgical procedure, preoperative instructions, postoperative care guidelines, and common patient concerns. The video includes both visual animations and spoken explanations.
  Interventions: Behavioral: Multimedia Health Education

INTERVENTIONS:
Behavioral: Multimedia Health Education — A 10-minute multimedia video is provided to the intervention group during their final preoperative clinic visit. All participants receive standard verbal and printed education from the ophthalmologist. The video includes visual and auditory content on cataract surgery, preoperative instructions, postoperative care, and common concerns. Baseline data (T0) are collected before the intervention, including demographics, visual acuity, physiological indicators, BAI, and self-care knowledge. Follow-ups occur at T1 (surgery day), T2 (1 week postop), and T3 (1 month postop), assessing anxiety, physiology, vision, and self-care.
  Arms: Multimedia Education Group

SUMMARY:
This study aims to examine the effectiveness of multimedia health education in reducing preoperative anxiety and enhancing self-care awareness among patients undergoing outpatient cataract surgery. A randomized group design will be employed, in which participants will receive either standard preoperative education or a multimedia-based intervention covering surgical procedures, precautions, and postoperative care. Primary outcomes include levels of surgical anxiety, assessed using validated anxiety scales, and self-care knowledge evaluated through structured questionnaires. Findings are expected to inform the development of patient-centered educational strategies and enhance perioperative care quality in cataract surgery settings.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of multimedia health education in reducing preoperative anxiety and improving postoperative care awareness among patients undergoing outpatient cataract surgery. A total of 118 patients scheduled for cataract surgery at an ophthalmology outpatient clinic will be randomly assigned to either the control group or the intervention group.

All participants will receive standard verbal preoperative instructions from their physician. In addition, the intervention group will view a 10-minute multimedia video covering the surgical procedure, precautions, and postoperative care. Baseline data-including demographics, visual acuity, physiological anxiety indicators, the Beck Anxiety Inventory (BAI), and a cataract-specific self-care knowledge questionnaire-will be collected during the final preoperative clinic visit.

Outcome data will be collected at three time points: before surgery, one week after surgery, and one month after surgery. Primary outcomes include changes in anxiety levels and self-care knowledge; secondary outcomes include physiological responses during surgery and postoperative visual recovery. The results are expected to support the use of multimedia education to enhance patient preparedness and care quality in cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Diagnosed with cataract and scheduled for elective phacoemulsification with intraocular lens implantation (first-time surgery)
* Able to communicate in Mandarin or Taiwanese
* Blood glucose <250 mg/dL and HbA1c <8% if diabetic (assessed by attending physician)

Exclusion Criteria:

Diagnosed with dementia or psychiatric disorders

* History of previous cataract surgery
* Severe hearing impairment (certified disability without hearing aid)
* Systolic blood pressure >160 mmHg on the day of surgery
* Preoperative visual acuity less than 0.05
* Undergoing combined ocular procedures (e.g., vitrectomy) during cataract surgery
* Unable to use digital devices required for the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety levels measured by the Beck Anxiety Inventory (BAI) | Time Frame: Day 0 (baseline, preoperative clinic visit), Day of Surgery, 1 Week Postoperative, 1 Month Postoperative
  Participants will complete the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire used to assess the severity of anxiety symptoms. The total score ranges from 0 to 63, with higher scores indicating greater levels of anxiety. Specifically, scores from 0-7 suggest minimal anxiety, 8-15 mild anxiety, 16-25 moderate anxiety, and 26-63 severe anxiety. The BAI will be administered at baseline and at three follow-up points.
Change in self-care knowledge related to cataract surgery | Time Frame: Day 0 (baseline, preoperative clinic visit), Day of Surgery, 1 Week Postoperative, 1 Month Postoperative
  Participants will complete a structured questionnaire designed to evaluate their knowledge of postoperative cataract care. Scores will be compared across time points to determine the impact of multimedia education.

SECONDARY OUTCOMES:
Change in heart rate | Time Frame: Day 0 (baseline, preoperative clinic visit), Day of Surgery
  Physiological indicators such as heart rate will be collected at designated time points to objectively assess anxiety responses.
Change in visual acuity following cataract surgery | Time Frame: Day 0 (baseline, preoperative clinic visit), 1 Week Postoperative, 1 Month Postoperative
  Visual acuity will be measured using a standard eye chart at follow-up to assess postoperative recovery.
Change in blood pressure | Day 0 (baseline, preoperative clinic visit), Day of Surgery
  Systolic and diastolic blood pressure (mmHg) will be recorded at baseline and on the day of surgery as objective physiological indicators of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Operating Room, Keelung, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu X, Vargas J, Green PHR, Bhagat G. Innate Lymphoid Cells and Celiac Disease: Current Perspective. Cell Mol Gastroenterol Hepatol. 2021;11(3):803-814. doi: 10.1016/j.jcmgh.2020.12.002. Epub 2020 Dec 10. PMID 33309944
- [Background] Jafarzadeh M, Saatchi M, Jafarnejadi P, Gooran M. Digital Radiographic Evaluation of the Quality of Different Root Canal Obturation Techniques in Deciduous Mandibular Molars after Preparation with Rotary Technique. J Dent (Shiraz). 2019 Sep;20(3):152-158. doi: 10.30476/DENTJODS.2019.44902. PMID 31579688